CLINICAL TRIAL: NCT01424241
Title: Metabolic, Cardiovascular and Body Composition Effects of Sandostatin LAR® Therapy of Acromegaly, Effect of Reduction of Serum Insulin-like Growth Factor 1 (IGF-1) Levels Into a New Normative Range
Brief Title: Effects of Sandostatin LAR® in Acromegaly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Pamela U. Freda, Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAC0246; CSMS995BUS57 (Other Grant/Funding Number: Novartis Pharmaceutical, Inc./Investigator Initiated study)
Record Dates: First submitted 2011-08-19; First posted 2011-08-26 (Estimated); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Acromegaly
Keywords: Sandostatin LAR
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sandostatin LAR (Experimental): Nine months of open label dose escalation Sandostatin LAR therapy.
  Interventions: Drug: Sandostatin LAR

INTERVENTIONS:
Drug: Sandostatin LAR — Open label dose escalation of Sandostatin LAR 10 mg, 20 mg, 30 mg, up to 40 mg if necessary.

SUMMARY:
This study aims primarily to determine the effect Insulin-like Growth Factor 1 (IGF-1) normalization into current IGF-I normal ranges with Sandostatin LAR® therapy on biochemical metabolic, cardiovascular and body composition parameters in patients with active acromegaly.

DETAILED DESCRIPTION:
A major goal of treatment of acromegaly is to normalize serum IGF-1 levels. Recently developed new normative data for serum IGF-1 levels has lowered the upper limit of normal for this hormone level. Octreotide, an analog of somatostatin, a synthetic form of the hypothalamic hormone somatostatin, which inhibits growth hormone (GH) release by blocking somatostatin receptors in the pituitary and on the tumor, is now available in a long acting depot formulation, Sandostatin LAR, that suppresses tumoral GH secretion and normalizes GH and IGF-1 levels in about 60% of patients. Although sandostatin LAR is Food and Drug Administration (FDA) approved for the therapy of acromegaly and is used clinically, its efficacy with respect to new normative IGF-1 ranges has not been studied. In addition, an important goal of therapy of acromegaly is to treat co-morbidities of the disease such as insulin resistance, which is common in acromegaly. Other important morbidities in acromegaly are hypertension and cardiovascular disease such as left ventricular hypertrophy (LVH). In this study the investigators will assess the effect of LAR therapy on biochemical parameters as well as important clinical endpoints of therapy of acromegaly.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age > 18 years) with diagnosis of Acromegaly ( previously confirmed by an elevated IGF-1 level)
2. IGF-1 concentrations> 10% above the upper limit of normal at screening
3. If the patient have undergone surgical resection of a pituitary adenoma, A minimum of two months must have elapsed post surgery prior to enrollment
4. May have a history of radiotherapy
5. Stable pituitary hormone supplements(x months) prior to baseline visit
6. if female ,

   1. not pregnant (as evidence by negative serum pregnancy test) or lactating; and
   2. If childbearing potential, agree to use a medically acceptable form of contraception (such as oral, implantable, or barrier contraception) from the screening, for the duration of the study, and for at least on month after study discontinuation or completion. Childbearing potential is defined as women who are not surgically sterile or not at least one year postmenopausal.
7. Sign and date an consent form document indicating that the subject (or legally acceptable representative) has been informed of and agrees to all pertinent aspects of trial

Exclusion Criteria:

1. Have other conditions that may result in abnormal growth hormone (GH) and/or IGF-1 concentrations (e.g., severe hepatic disease, severe renal disease Malnutrition, treatment with levodopa)
2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 x Upper limit of normal or clinically significant hepatic disease
3. Prior somatostatin analog therapy within 6 months of the screening visit
4. Other medical therapy for acromegaly for 6 weeks to screening visit
5. Visual field defects or other neurological symptoms due to tumor mass
6. Have known or suspected drug or alcohol abuse
7. Have received an investigational medication within four week prior to screening or is scheduled to received any investigational medication during the study
8. Do not have ability to fully comprehend the nature of the study, to follow instructions, cooperate with study procedures, and/or are unable to adhere to the visit scheduled outlined in the protocol
9. Have other severe acute or chronic medical or psychiatry condition or Laboratory abnormality that may increase the risk associated with study Participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
10. Patient who have known hypersensitivity to Sandostatin acetate or other related drug or compound
11. Patient with current gallstones
12. Patient who have received supraphysiologic doses of glucocorticoid within the past 6 months (except for peri-operative (<3 days duration) of dexamethasone) or who currently received chemotherapeutics agents, or exogenous growth hormone
13. Patients who have received other investigational drugs administered or Received within 30 days of study entry
14. Patients who exhibit symptoms indicative of intolerance during the 2 weeks Course of Sandostatin injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-10; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela U Freda, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Dose Escalation Study of Sandostatin LAR Therapy: Acromegaly is a rare disorder due in almost all cases to a GH secreting tumor of the pituitary gland. The initial treatment is typically surgical removal of the tumor, but after this many patients have residual disease requiring additional therapy. For most patients this therapy is medical with a somatostatin analog.
  In addition to biochemical control, important and often overlooked goals of acromegaly care are to treat its associated co-morbidities in particular insulin resistance and diabetes mellitus, hypertension and cardiovascular (CV) disease. Changes in body composition in acromegaly may be integral to the development of insulin resistance and increased CV risk.
  Therefore, this study sought to examine the effect of lowering of serum IGF-I levels into the current more stringent normal range during treatment with octreotide LAR on metabolic parameters, body composition and cardiovascular risk profile in patients with acromegaly.
Period: Overall Study
Arm/Group | Open Label Dose Escalation Study of Sandostatin LAR Therapy
Started | 21
Completed | 18
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Time constraints | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Dose Escalation Study of Sandostatin LAR Therapy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 44.9 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 21
IGF-1 Level [Mean (Full Range); unit: ng/ml] | 336 [287 to 385]

OUTCOME MEASURES:

1. Primary Outcome: IGF-1 Level on Sandostatin LAR
Description: Mean IGF-1 level on treatment with Sandostatin LAR in whole population and responders (normal IGF1) and non responders(elevated IGF-1)
Time Frame: Up to 9 months
Population: This study was open to adult patients with active acromegaly, either newly diagnosed or failing other therapies who met the following inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Open Label Dose Escalation of Sandostatin LAR Therapy: The study population is limited to patients with acromegaly presenting to the Neuroendocrine Unit.
- Responders: Normal IGF-1 Group
- Non Responders: Elevated IGF-1 Group
Arm/Group | Open Label Dose Escalation of Sandostatin LAR Therapy | Responders | Non Responders
Number analyzed (Participants) | 18 | 10 | 8
ng/mL | 336 (209) | 186 (42.4) | 487 (200.4)
Statistical Analysis 1: Comparison: Open Label Dose Escalation of Sandostatin LAR Therapy; None available; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 300
Statistical Analysis 2: Comparison: Responders vs Non Responders; Test type: Superiority; p < .05, t-test, 2 sided; Mean Difference (Final Values) = 1.6

2. Secondary Outcome: Cardiovascular Risk Markers on Sandostatin LAR: C-reactive Protein (CRP) Levels
Description: Levels of C-reactive protein (CRP) in whole study group, responders (normal IGF-1) and non responders (elevated IGF-1) groups. Higher values are a worse outcome.
Time Frame: Up to 9 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Open Label Dose Escalation of Sandostatin LAR Therapy | Responders | Non Responders
Number analyzed (Participants) | 18 | 10 | 8
mg/L | 2.05 (3.5) | 2.89 (4.79) | 1.21 (1.2)

3. Secondary Outcome: Cardiovascular Risk Markers on Sandostatin LAR: Homocysteine Levels
Description: Levels of homocysteine in whole study group, responders (normal IGF-1) and non responders (elevated IGF-1) groups. Higher values are a worse outcome.
Time Frame: Up to 9 months
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Open Label Dose Escalation of Sandostatin LAR Therapy | Responders | Non Responders
Number analyzed (Participants) | 18 | 10 | 8
µmol/L | 9.98 (5.8) | 10.57 (5.56) | 9.40 (6.4)

4. Secondary Outcome: Cardiovascular Risk Markers on Sandostatin LAR: Lipid Levels
Description: Levels of lipid panel (cholesterol, triglycerides, and Lipoprotein A) in whole study group, responders (normal IGF-1) and non responders (elevated IGF-1) groups. Higher values are a worse outcome.
Time Frame: Up to 9 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Label Dose Escalation of Sandostatin LAR Therapy | Responders | Non Responders
Number analyzed (Participants) | 18 | 10 | 8
mg/dL
  Total cholesterol | 173.75 (42.9) | 182.44 (49.78) | 162.57 (32.1)
  LDL cholesterol | 101.56 (40.7) | 108.7 (45.38) | 92.43 (34.9)
  HDL Cholesterol | 52.17 (14.6) | 53.44 (16.19) | 50.89 (13.6)
  Triglycerides | 95.2 (36.2) | 88.38 (38.13) | 103 (35.1)
  Lipoprotein a | 55.31 (68.9) | 71.45 (85.95) | 34.56 (33.4)

ADVERSE EVENTS:
Arm/Group | Open Label Dose Escalation Study of Sandostatin LAR Therapy
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes